CLINICAL TRIAL: NCT00491907
Title: Effect of Folic Acid on Endothelial and Baroreceptor Function in Patients With Heart Failure
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: recruitment is finished
Sponsor: University of Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FolicAcid881
Record Dates: First submitted 2007-06-25; First posted 2007-06-26 (Estimated); Last update posted 2007-10-02 (Estimated); Status verified 2007-10

CONDITIONS: Heart Failure
Keywords: folic acid; endothelial function; baroreceptor function; heart failure
MeSH Terms: conditions — Heart Failure | interventions — Folic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: folic acid 5mg/day

SUMMARY:
The randomized, double-blind, placebo-controlled study aim to evaluate the effect of 1-month therapy with folic acid (5 mg/day) on endothelial function and baroreceptor function in patients with heart failure.

Endothelial function will be studied non-invasively with flow-mediated dilation while for eveluating baroreceptor function sympathetic nervous system activity will be measured directly with microneurography in baseline condition and during infusion of sodium-nitroprusside.

DETAILED DESCRIPTION:
Endothelial and baroreceptor function are impaired in patients with heart failure.

Impaired baroreflex control of the heart and peripheral circulation and endothelial dysfunction are thought to play an important pathophysiological role in chronic heart failure and confers a poor prognosis.

In patients with essential hypertension we demonstrated an improvement in baroreceptor function after treatment with folic acid.

Therefore, the aim of the present randomized, double-blind, placebo-controlled study was to evaluate endothelial function and baroreceptor function in patients with heart failure before and after 1-month therapy with folic acid (5 mg) or placebo.

Endothelial function will be assessed with novel high-resolution ultrasound devices, which allows to investigate endothelial function in vivo. This method makes use of the property of the endothelium to release nitric oxide in response to shear stress and increased flow as previously described. Endothelium-dependent flow-mediated dilation (FMD) and endothelium-independent glycerol trinitrate (GTN) (0.4 mg sublingual, Nitrolingual Spray, Pohl-Boskamp, Germany)-induced vasodilation of the brachial artery will be assessed by a high-resolution ultrasound vessel wall tracking device with a 10 MHz linear array transducer . FMD of the brachial artery is induced by release of a wrist cuff inflated 50 mmHg above systolic pressure for 5 minutes. After sublingual GTN application, used as endothelium-independent stimulus, the diameter will be recorded every 30 seconds for 6 minutes.

Multifiber recordings of muscle sympathetic nerve activity will be obtained from the peroneal nerve posterior to the fibular head with tungsten microelectrodes. The sympathetic nervous activity will be measured continuously together with ECG, respiration rate and blood pressure. Baroreceptor modulation of muscle sympathetic nerve activity and heart rate would be assessed by intravenous infusion of sodium nitroprusside.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure (min. NYHA ll, LVEF <50%)
* Not smokers
* Written informed consent

Exclusion Criteria:

* Unstable heart failure
* Smoking
* Unstabile Angina Pectoris
* Endocrinologic disease such as Diabetes mellitus, Hypo- und Hyperthyroidism
* Alcohol abuse
* Epilepsia
* Treatment with folic acid antaponists Trimethoprim, Pyrimethamin, Methotrexat..
* Participation to one other clinical Study within 1 Month

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-10; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
change in endothelial function | 1 month
change in baroreceptor function | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Georg Noll, MD, Principal Investigator — Cardiovascular Center, University Hospital Zurich, Zurich, Switzerland